CLINICAL TRIAL: NCT07195279
Title: Psychometric and Physiological Assessment of the Effects of Vir-tual Reality in Cardiovascular Rehabilitation: a Randomized Con-trolled Trial
Brief Title: Psychometric and Physiological Assessment of the Effects of Vir-tual Reality in Cardiovascular Rehabilitation
Acronym: VRHEART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.R.C.C.S. Fondazione Santa Lucia (Other)
Collaborators: University of Roma La Sapienza (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FSLVRHEART
Record Dates: First submitted 2025-09-01; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Cardiac Rehabilitation
Keywords: Virtual Reality; Rehabilitation; Cardiac Rehabilitation
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Model Description
Who Masked: Investigator, Outcomes Assessor
Masking Description: Masking Description
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (calisthenics sessions) (Active Comparator): The control group of this study performed a conventional cardiac rehabilitation protocol that consisted of 1.5 hour group calisthenics sessions with a 10-minute break, held six times per week. This was accompanied by aerobic reconditioning exercises on a stationary bike or treadmill, depending on medical prescription and the patient's health status.
  Interventions: Other: Control Group
- Experimental Group (VR experience) (Experimental): The VR intervention consisted of a simulated driving experience delivered over nine sessions, three times per week, each lasting 20 minutes, over a three-week period. Patients were exposed to diverse driving scenarios, specifically: urban streets (featuring intersections, traffic lights, and pedestrians to simulate complex urban environments), ring roads (designed for practicing smooth and confident high-speed driving in dense traffic), and tunnels (sections aimed at gradually desensitizing users to claustrophobic responses during driving).
  Interventions: Other: Experimental Group

INTERVENTIONS:
Other: Experimental Group — The VR intervention consisted of a simulated driving experience delivered over nine sessions, three times per week, each lasting 20 minutes, over a three-week period. The virtual reality (VR) therapy employed a full immersion approach, delivering intense multisensory visual-auditory stimulation. Patients were exposed to diverse driving scenarios, specifically: urban streets (featuring intersections, traffic lights, and pedestrians to simulate complex urban environments), ring roads (designed for practicing smooth and confident high-speed driving in dense traffic), and tunnels (sections aimed at gradually desensitizing users to claustrophobic responses during driving).
  Arms: Experimental Group (VR experience)
Other: Control Group — Conventional cardiac rehabilitation protocol consisted of 1.5-hour group calisthenics sessions with a 10-minute break, held six times per week. This was accompanied by aerobic reconditioning exercises on a stationary bike or treadmill, depending on medical prescription and the patient's health status.
  Arms: Control Group (calisthenics sessions)

SUMMARY:
Virtual reality (VR) is a high-end user-computer interface involving real-time stimulation and interaction of an embedded subject through visual and auditory sensorial channels, based on a synthetic environment in which the subject feels to be present. Over the past few decades, VR has been extensively used in psychological and neuroscientific research, as well as clinical applications, yielding promising results for diverse clinical conditions. Furthermore, VR has also been employed in the cardiovascular field across various settings, including cardiac rehabilitation, interventional cardiology, and cardiac surgery, to assess both physiological and psychological outcomes.

The benefits of using VR may stem from its ability to be customized, potentially enhancing the rehabilitation experience by offering cognitive, emotional, and physical advantages. It can improve patients' motivation and engagement, reduce anxiety. In general, in the context of cardiac rehabilitation, the impact of VR appears to be more closely linked to improvements in mental health, particularly in relation to psychological aspects such as mood enhancement, stress reduction, and increased emotional well-being. These benefits may be due to the immersive and engaging nature of VR, which can provide a sense of novelty, distraction from discomfort, and a greater feeling of control over the rehabilitation process. However, current evidence does not clearly demonstrate its superiority over conventional approaches in other important outcomes, including treatment adherence, patient satisfaction, and overall quality of life. The aim of this study was to test the efficacy of integrating the use of a VR system based on driving simulation in cardiac rehabilitation through a randomized controlled trial.

DETAILED DESCRIPTION:
The study is an RCT. The control group of this study performed a conventional cardiac rehabilitation protocol that consisted of a 1.5-hour group calisthenics sessions with a 10-minute break, held six times per week.

Patients were randomly allocated to the experimental virtual reality group and underwent the standard cardiac rehabilitation program, but some sessions were substituted by the virtual reality rehabilitation protocol. The VR intervention consisted of a simulated driving experience delivered over nine sessions, three times per week, each lasting 20 minutes, over a three-week period. Participants observed the virtual scenario through Meta Quest 2 head-mounted display. The 3D environment consisted of a realistic 3D model of a car's interior, simulating the driver's perspective (1:1 scale). The virtual cockpit incorporated an interactive steering wheel, controlled by participants from their perspective using Meta Controllers. This interaction, however, did not alter the vehicle's movement path. To optimize immersion, the Meta Controllers were rendered as hands, integrated with a 3D avatar model. The various scenarios the patient encountered corresponded to a progressively increasing level of difficulty as the rehabiltative sessions proceeded. Examples of challenging elements included narrow roads, urban traffic, tunnel driving, and high-speed roads. Each session lasted approximately 20 minutes, which was the time required to complete the driving route. However, the session might end earlier if the patient was unable to continue.

ELIGIBILITY:
* Diagnosis of cardiovascular disease and need for intensive inpatient cardiac rehabilitation after cardiac surgery;
* Age over 18 years;
* Absence of comorbidities (cognitive deficits, psychiatric syndromes, visual sensitivity; physical conditions);
* Ability to understand and follow instructions provided by physiotherapists.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-01-07 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Emotional benefit and distress reduction | This scale was administered at three time points: as baseline, before the beginning of intervention (Day 0), after the first session of treatment (Day 1) and after intervention completion (Day 21)
  Hospital Anxiety and Depression Scale (HADS): A 14-item scale used to assess anxiety (7 items) and depression (7 items) levels related to illness. This scale is widely used to assess general mental health in hospitalized patients and chronically ill patients, allowing for symptom monitoring rather than making a specific diagnosis.

SECONDARY OUTCOMES:
Upper limb Range of Motion | This evaluation was made at two time points: after the first session of treatment (Day 1) and after intervention completion (Day 21)
  Assessment of changes in upper limb range of motion: shoulder flexion/extension, elbow flexion/extension.

OTHER OUTCOMES:
Physiological exertion | This evaluation was made on: Day 1, Day 3, Day 5, Day 9, Day 11, Day 13, Day 17, Day 19, Day 21
  Physiological evaluation of stress induced by VR was measured collecting heart rate variability, as the number of R-R intervals in the timeframe of one second.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Iosa, PhD, Associate Professor, Principal Investigator — IRRCS Santa Lucia foundation
Locations (1):
- IRCCS Santa Lucia foundationa and Nomentana Hospital, Rome, Lazio, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be available under request to corresponding Author after publications